CLINICAL TRIAL: NCT02204865
Title: Sleep-Disordered Breathing in Patients With Implanted Cardiac Devices: Validation of the ApneaScan Algorithm and Implications for Prognosis
Brief Title: Validation of the ApneaScan Algorithm in Sleep Disordered Breathing
Acronym: ApneaScan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 14/LO/0077
Record Dates: First submitted 2014-04-11; First posted 2014-07-30 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Sleep-Disordered Breathing; Heart Failure
Keywords: Sleep-Disordered Breathing; Sleep Apnoea; Heart failure
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure | interventions — Device Lead Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker/ICD with ApneaScan: Patients with HFREF due to receive a pacemaker or ICD with ApneaScan function
  Interventions: Device: Pacemaker/ICD

INTERVENTIONS:
Device: Pacemaker/ICD — Implantation of an ICD or CRT device with ApneaScan function
  Other Names: Invive, Inliven, Incepta, Energen, Autogen devices.

SUMMARY:
Sleep disordered breathing, in which patients my breath deeply, shallowly or stop breathing for periods whilst asleep, is common in heart failure and associated with a poor prognosis. This study aims to validate a novel function available on certain pacemakers which is designed to detect this condition.The investigators hypothesize that ApneaScan can accurately detect moderate to severe sleep disordered breathing in patients with heart failure as compared against an Embletta sleep study. The investigators will also follow up our patients for 2 years to determine whether the severity of sleep disordered breathing as assessed by ApneaScan correlates with prognosis.

DETAILED DESCRIPTION:
72 patients with heart failure with reduced ejection fraction (HFREF) who have been selected to receive an Implantable Cardioverter-Defibrillator (ICD) or Cardiac Resynchronization Therapy Pacemaker or Defibrillator (CRT-P/D) will undergo pre-implant assessment with an echocardiogram, B-type Natriuretic Peptide (BNP) level, 6 minute walk test, Minnesota living with heart failure and Epworth sleepiness questionnaires. The patients will then have the device implanted. 6 to 8 weeks later the patent will undergo an Embletta home sleep study and download of the ApneaScan data from the device. The mean Apnoea-Hypopnoea Index (AHI) from the ApneaScan download will be compared with that derived from the sleep study. The patients will also have a repeat 6 minute walk test, echocardiogram and BNP level.

2 years after device implantation, all patients will be followed up to document deaths, hospital admissions, Atrial Fibrillation (AF) burden and appropriate therapies from ICD devices.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with reduced ejection fraction (EF < 40%)
* Due to receive a device with ApneaScan function
* Able to give informed consent
* Ambulatory

Exclusion Criteria:

* Known sleep disordered breathing on Non-Invasive Ventilation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure with reduced ejection fraction (EF <40%) due to receive a Boston Scientific ICD/CRTD/P with ApneaScan function.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The Apnoeic-Hypopnoeic Index (AHI) | 18 months
  We will compare that AHI from the ApneaScan pacemaker algorithm against the AHI from an Embletta sleep study.

SECONDARY OUTCOMES:
Adverse heart failure events | 2 years
  Comprising hospital admissions for heart failure, AF burden, VF and VT burden and mortality

OTHER OUTCOMES:
B-Type Natriuretic peptide (BNP) concentration | 2 years
  BNP concentration correlated with severity of SDB
Ejection fraction on echocardiography | 2 years
  Correlation of ejection fraction and severity of SDB
6 minute walk test distance | 2 years
  Correlation between 6MWTd and severity of SDB

CONTACTS AND LOCATIONS:
Overall Officials: Ali Vazir, PhD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Trust, London, London, United Kingdom